CLINICAL TRIAL: NCT01823068
Title: A Phase II Study of Vandetanib in Patients With Non-small Cell Lung Cancer Harboring RET Rearrangement
Brief Title: Vandetanib in Advanced NSCLC With RET Rearrangement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Se-Hoon Lee, Associate Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-09-089-01
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung cancer; RET fusion; Vandetanib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib treatment arm (Experimental): Vandetanib 300 mg once daily orally
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — Patients will begin on once daily vandetanib at 300 mg with one cycle of 4 weeks.
  Other Names: Caprelsa

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of vandetanib, in patients with advanced non-small-cell lung cancer harboring RET gene rearrangement. In 2011, gene rearrangement between RET and KIF5B gene (fusion) was discovered in a young, male lung cancer patient. The following studies showed that this gene rearrangement was critical for tumor initiation and maintenance. Of note, the growth and signaling properties mediated by KIF5B-RET were diminished after treatment with vandetanib.

Until now, RET rearrangements have been known in thyroid cancers. Vandetanib, a multi-kinase inhibitors with anti-RET activity, is an FDA-approved drug for the treatments of adults with metastatic medullary thyroid cancers who are ineligible for surgery and who have progressive or symptomatic disease. This study aimed to examine the efficacy and safety of this drug, for the treatment of advanced lung cancer harboring RET rearrangement.

DETAILED DESCRIPTION:
Patients will be screened so as to confirm RET fusion in their tumor tissue. RET fusion will be tested using fluorescence in situ hybridization (FISH) at central laboratory. Central laboratory of this study is the department of pathology at Seoul National University Hospital (SNUH) and tumor specimen should be sent to department of pathology at SNUH. Only patients whose tumor have confirmed RET gene fusion are eligible for this study.

Enrolled patients will begin on once daily vandetanib at 300 mg with one cycle of 4 weeks. Renal-impaired patients (defined as patients with creatinine clearance ≥30 to <50 mL/min at screening) will start treatment at the lower dose of 200 mg. Treatment will be continued till progression, unacceptable toxicity, or till 1 year. Vandetanib can be administered after 1 year to the patients with benefit from vandetanib.

During the administration of vandetanib, vital signs, physical examination, ECOG performance status, height, weight, hematology and chemistry test, ECG, adverse events and concomitant drugs will be evaluated every four weeks (one cycle, for the first 6 months) or eight weeks (two cycles, from 6 months to 1 year) and, if necessary, chest X-ray and pregnancy test will also be performed. CT for tumor assessment will be performed once every 8 weeks for 1 year. If the disease progression is suspected, the test can be additionally conducted at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Female or male aged 18 years or over
* Histologically confirmed locally advanced or metastatic (stage IIIB or IV) NSCLC
* Failure after platinum-based chemotherapy
* Presence of a RET fusion in an archival or newly acquired NSCLC tumor specimen (RET fusion should be performed in central laboratory by FISH)
* ECOG performance status of 0, 1 or 2
* Negative pregnancy test (urine or serum) for female patients of childbearing potential
* Measurable disease according to RECIST 1.1 criteria
* Life expectancy of >12 weeks
* Able to swallow study medication
* If the subject is on the course of radiotherapy, one can be enrolled after radiotherapy

Exclusion Criteria:

* Involvement in the planning/conduct of this study
* Previous enrollment in the present study
* Previous exposure to vandetanib
* Unstable brain metastases or spinal cord compression that requires treatment (The patients with treated brain metastases who are on a stable dose of steroids can be included)
* Major surgery within 28 days before starting treatment
* The last dose of prior chemotherapy received less than 28 days prior to starting treatment
* Any unresolved chronic toxicity greater than CTCAE grade 2 from previous anticancer therapy
* Serum bilirubin greater than 1.5 x the upper limit of reference range (ULRR)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) greater than 2.5 x ULRR, or greater than 5.0 x ULRR if judged by the investigator to be related to liver metastases
* Creatinine clearance <30 mL/min (Patients with moderate renal impairment defined as screening creatinine clearance ≥30 to <50 mL/min will start vandetanib at a reduced dose of 200 mg once daily and will continue this dose throughout the study, unless further dose reduction is required)
* Unacceptable electrolyte imbalance (Potassium <4.0 mmol/L despite supplementation, Magnesium below normal range despite supplementation, Calcium as evaluated by either ionized or standard serum tests: ionized calcium below the normal range or serum calcium above the CTCAE grade I upper limit)
* Significant cardiac event (e.g. myocardial infarction), superior vena cava syndrome, NYHA classification of heart disease ≥2 within 12 weeks before starting treatment, or presence of cardiac disease that in the opinion of the investigator increases the risk of ventricular arrhythmia
* History of ventricular arrhythmia, which is symptomatic or requires treatment (CTCAE grade 3), symptomatic or uncontrolled atrial fibrillation, or asymptomatic sustained ventricular tachycardia. (Patients with atrial fibrillation controlled by medication are permitted)
* Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure > 100 mmHg)
* Past medical history of, or clinically active interstitial lung disease
* Evidence of severe or uncontrolled systemic disease
* Previous or current malignancies of other histologies within the last 3 years. (In situ carcinoma of the cervix, adequately treated basal cell or squamous cell carcinoma of the skin is exceptionally permitted)
* Congenital long QT syndrome
* Any concomitant medications that are known to be associated with Torsades de Pointes or potent inducers of cytochrome P450 3A4 (CYP3A4) function and/or any prohibited medications
* History of QT prolongation associated with other medication that required discontinuation of that medication
* QTcB correction unmeasurable or >480 ms on screening ECG
* Participation in a clinical study and/or receipt of an investigational drug within 28 days prior to enrollment
* Females only - currently pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2014-12-29 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR will be evaluated through the frequency analysis with 95% confidence interval.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  PFS will be examined with Kaplan-Meier method.
Disease-control rate (DCR) | 1 year
  DCR will be evaluated through the frequency analysis with 95% confidence interval.
Overall survival (OS) | 2 years
  OS will be examined with Kaplan-Meier method.
Number of Participants with Adverse Events | 1 years
  Regarding safety endpoints, all adverse events will be individually graded based on the CTCAE version 4.03. The number of participants with adverse events will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Background] Ju YS, Lee WC, Shin JY, Lee S, Bleazard T, Won JK, Kim YT, Kim JI, Kang JH, Seo JS. A transforming KIF5B and RET gene fusion in lung adenocarcinoma revealed from whole-genome and transcriptome sequencing. Genome Res. 2012 Mar;22(3):436-45. doi: 10.1101/gr.133645.111. Epub 2011 Dec 22. PMID 22194472
- [Background] Takeuchi K, Soda M, Togashi Y, Suzuki R, Sakata S, Hatano S, Asaka R, Hamanaka W, Ninomiya H, Uehara H, Lim Choi Y, Satoh Y, Okumura S, Nakagawa K, Mano H, Ishikawa Y. RET, ROS1 and ALK fusions in lung cancer. Nat Med. 2012 Feb 12;18(3):378-81. doi: 10.1038/nm.2658. PMID 22327623
- [Background] Lipson D, Capelletti M, Yelensky R, Otto G, Parker A, Jarosz M, Curran JA, Balasubramanian S, Bloom T, Brennan KW, Donahue A, Downing SR, Frampton GM, Garcia L, Juhn F, Mitchell KC, White E, White J, Zwirko Z, Peretz T, Nechushtan H, Soussan-Gutman L, Kim J, Sasaki H, Kim HR, Park SI, Ercan D, Sheehan CE, Ross JS, Cronin MT, Janne PA, Stephens PJ. Identification of new ALK and RET gene fusions from colorectal and lung cancer biopsies. Nat Med. 2012 Feb 12;18(3):382-4. doi: 10.1038/nm.2673. PMID 22327622
- [Background] Gautschi O, Zander T, Keller FA, Strobel K, Hirschmann A, Aebi S, Diebold J. A patient with lung adenocarcinoma and RET fusion treated with vandetanib. J Thorac Oncol. 2013 May;8(5):e43-4. doi: 10.1097/JTO.0b013e31828a4d07. No abstract available. PMID 23584301
- [Background] Falchook GS, Ordonez NG, Bastida CC, Stephens PJ, Miller VA, Gaido L, Jackson T, Karp DD. Effect of the RET Inhibitor Vandetanib in a Patient With RET Fusion-Positive Metastatic Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 May 20;34(15):e141-4. doi: 10.1200/JCO.2013.50.5016. Epub 2014 Nov 3. No abstract available. PMID 25366691
- [Derived] Lee SH, Lee JK, Ahn MJ, Kim DW, Sun JM, Keam B, Kim TM, Heo DS, Ahn JS, Choi YL, Min HS, Jeon YK, Park K. Vandetanib in pretreated patients with advanced non-small cell lung cancer-harboring RET rearrangement: a phase II clinical trial. Ann Oncol. 2017 Feb 1;28(2):292-297. doi: 10.1093/annonc/mdw559. PMID 27803005
- [Derived] Wu H, Shih JY, Yang JC. Rapid Response to Sunitinib in a Patient with Lung Adenocarcinoma Harboring KIF5B-RET Fusion Gene. J Thorac Oncol. 2015 Sep;10(9):e95-e96. doi: 10.1097/JTO.0000000000000611. No abstract available. PMID 26291023